CLINICAL TRIAL: NCT06016699
Title: Effect of Protons Versus Photons on Immunological Function in Head and Neck Cancer: a Pilot Study
Brief Title: Immunological Function After Radiation With Either Proton or Photon Therapy
Acronym: PRO-IMMUNO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: NL75013.042.20
Record Dates: First submitted 2023-08-23; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: HNSCC; Head and Neck Cancer; Oropharynx Cancer; Hypopharynx Cancer; Larynx Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Chemoradiation with protons: HNSCC patients treated with standard-of-care chemoradiation with protons.
  Interventions: Other: blood draws
- Chemoradiation with photons: HNSCC patients treated with standard-of-care chemoradiation with photons.
  Interventions: Other: blood draws
- Radiation with protons: HNSCC patients treated with standard-of-care radiation with protons.
  Interventions: Other: blood draws
- Radiation with photons: HNSCC patients treated with standard-of-care radiation with photons.
  Interventions: Other: blood draws

INTERVENTIONS:
Other: blood draws — Blood draws to collect PBMCs at baseline (week 0), during (chemo)radiation treatment (end of week 3 and/or before delivery of cycle 4 of cisplatin) and after conclusion of (chemo)radiation (week 9, week 12, week 20, week 34 and week 60, respectively 1 week, 5 weeks, 3 months, 6 months and 12 months after completion of (chemo)radiation) in order to compare immunological function upon treatment with either protons or photons

SUMMARY:
This is a pilot prospective observational cohort study, comprising patients with head and neck cancer (HNSCC) treated with standard of care definitive (chemo)radiation either with photons or protons. Patients will be assigned for protons or photons based on the guidelines of the National Indication Protocol for Proton therapy of the Netherlands.

Immunological function will be evaluated by the collection of peripheral blood mononuclear cells (PBMCs). Blood samples will be collected at baseline, during (chemo)radiation (end of week 3 and/or before week 4 of treatment) and after completion of (chemo)radiation (week 9, week 12, week 20, week 34 and week 60, respectively 1 week, 5 weeks, 3 months, 6 months and 12 months after completion of (chemo)radiation). To quantify immunological function, PBMCs collected during (chemo)radiation and after (chemo)radiation will be compared with that before (chemo)radiation (week 0), using IFN-γ-ELISPOT to screen for the presence of antigen-specific T-cell responses. Furthermore, flow cytometry panels will be used to determine global changes in immune cell proficiency.

Histological evaluation will take place at baseline and week 3 to examine changes in immune infiltration within tumour tissue during proton versus photon (chemo)radiation. This biopsy part of the study is optional for the patient. Archival tissue from the biopsy that was taken at diagnosis will be used for the baseline assessments. Biopsy at week 3 week will be taken for all patients who agree to participate in this optional part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed stage III-IV HNSCC of the oral cavity, oropharynx, hypopharynx or larynx.
* Treatment with definitive (chemo)radiation (70 Gy with or without weekly cisplatin) with photons or protons.
* Age of 18 years and older.
* Elective or therapeutic bilateral neck irradiation indicated.
* Written informed consent according to local guidelines.

Exclusion Criteria:

* Unilateral radiotherapy of the neck.
* (Diagnostic) resection of the primary tumour.
* Chemoradiation with carboplatin and 5-FU or radiation combined with cetuximab.
* History of an autoimmune disease or other systemic intercurrent disease that might affect the immunocompetence of the patient, or current or prior use (4 weeks before start of the trial) of high dose immunosuppressive therapy.
* Additional malignancy that is progressing or has required active treatment within the past 3 years. Note: participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Participation in a study of an investigational agent or has used an investigational device within 4 weeks prior enrolment in this trial. Note: participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
* Active infection requiring systemic therapy.
* Current pregnancy.
* History or current evidence of any condition, therapy or laboratory abnormality that might confound the results of this trial, interfere with the subject's participation for the full duration of this trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited at the Univeristy Medical Center Groningen (UMCG( and consists of adult patients recently diagnosed with stage III-IV HNSCC. Both photon and proton radiation are standard-of-care treatments for patients with HNSCC.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
The difference in antigen-specific immunity in HNSCC patients undergoing (chemo)radiation with protons versus photons. | At baseline (week 0), during (chemo)radiation (week 3) and after (chemo)radiation (week 9, week 12, week 20, week 34 and week 60, respectively week, 5 weeks, 3 months, 6 months and 12 months after completion of (chemo)radiation)
  Antigen-specific immunity will be assessed by monitoring antigen-specific T-cell responses in peripheral blood before, during and after (chemo)radiation (up to 12 months after completion of (chemo)radiation) to viral peptides such as SARS-CoV-2 peptides and CEF peptides (CMV, EBV and Influenza).

SECONDARY OUTCOMES:
Differences in composition and function of circulating immune cells during and after (chemo)radiation with protons versus photons. | At baseline (week 0), during (chemo)radiation (week 3) and after (chemo)radiation (week 9, week 12, week 20, week 34 and week 60, respectively week, 5 weeks, 3 months, 6 months and 12 months after completion of (chemo)radiation)
  Differences in composition and function of circulating immune cells will be determined by flow cytometry-based assays using marker for e.g. T- and B-lymphocytes and different myeloid cells such as derived suppressor cells.
Immune infiltrate composition within the primary tumour tissue before and during (chemo)radiation with photons versus protons (optional part of the study). | At baseline (week 0) and during (chemo)radiation (week 3)
  Immunohistological staining will be performed on these tumour tissues to assess changes in the composition of immune cells after (chemo)radiation with protons versus photons These assays include molecular analyses and immunohistochemical staining to characterize the type of the intratumoral immune cell infiltrate. In particular, immunohistochemical staining to identify immune cell populations and T cell subpopulations within the tumour tissue can be applied, including, but not limited to, CD4, CD8, FoxP3, CD20, CD163, CD68, PDL1 and PD1. Both changes in absolute numbers and ratios of different immune cell types will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen (UMCG), Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided